CLINICAL TRIAL: NCT05889780
Title: Screening for and Responding to Food Insecurity Among Simmons Infusion Patients at RedBird
Brief Title: Screening for and Responding to Food Insecurity Among Infusion Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kelseanna Hollis-Hansen, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 48557
Record Dates: First submitted 2023-05-18; First posted 2023-06-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Diet, Healthy; Nutrition, Healthy
Keywords: Food insecurity; Food pantry; Nutrition intervention
MeSH Terms: conditions — Neoplasms | interventions — Fast Foods

STUDY DESIGN:
Intervention Model Description: In the proposed study, infusion patients that screen positve for food insecurity that enroll in the study will be randomized to receive one of three evidence-based food security programs: 1) Pantry only - Referrals to an onsite food pantry or receipt of emergency food boxes if the onsite pantry is not open by 2024, 2) Pantry + nutritious no-prep, ready-to-eat meals, or 3) Pantry + $75 grocery vouchers for three-months.
Masking Description: It is not possible to mask staff or participants in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pantry only (Active Comparator): Referrals to onsite food pantry or emergency food boxes from partner pantry if onsite pantry is not open by 2024.
  Interventions: Other: Food pantry referrals
- Nutritious, no-prep meals (Experimental): Participants will receive up to 12 nutritious no-prep meals per month (three meals per week) for three-months.
  Interventions: Other: Food pantry referrals; Other: No-prep, ready-to-eat meals
- Vouchers (Experimental): Participants will receive $75 vouchers each month for three-months.
  Interventions: Other: Food pantry referrals; Other: Vouchers

INTERVENTIONS:
Other: Food pantry referrals — Clients receive food for up to 21 meals per person in the household each month.
Other: No-prep, ready-to-eat meals — 12 nutritious no-prep, ready-to-eat meals are provided each month.
  Arms: Nutritious, no-prep meals
Other: Vouchers — A $75 voucher is provided each month and participants are instructed to use the voucher to purchase food or transportation to food retailers.
  Arms: Vouchers

SUMMARY:
Food insecurity impacts 1 in 8 people in the United States and 1 in 4 people receiving cancer treatment. Food insecurity is associated with poor dietary quality, adverse health conditions (e.g., Type 2 diabetes, overweight and obesity, hypertension), and worse cancer treatment outcomes. To effectively address food insecurity among people with cancer, screening and effective response programs are needed.

The Food to Overcome Disparities (FOOD) program screens breast cancer patients for food insecurity and refers people who screen positive to 11 clinic pantries across New York City. In addition to clinic referrals, researchers have found the addition of monthly grocery vouchers or home grocery delivery to be even more effective at improving treatment completion rates than pantry access alone. Another innovative food security strategy, nutritious no-prep, ready-to-eat meals may also be helpful for patients given that no-prep meals reduce the time and physical demand of food preparation.

Nutritious no-prep, ready-to-eat meals have been positively associated with improvements in healthy eating index (HEI) scores, fewer instances of hypoglycemia, and improved quality of life among people with food insecurity that have diabetes, but has yet to be tested among patients with cancer. People receiving cancer treatment, such as infusion services, often report fatigue and other barriers to food preparation, which make no-prep, ready-to-eat meals another potential solution to cancer-specific challenges to healthy eating.

In the present study the investigators will test which evidence-based strategies are most effective and well-liked by patients and will inform the development of a comprehensive food security response program at the Harold C. Simmons Comprehensive Cancer Center.

DETAILED DESCRIPTION:
In the proposed study, the study team will screen infusion patients for food insecurity and refer those who screen positive to enroll in a randomized controlled trial where participants will receive one of three evidence-based food security programs: 1) Pantry only - Referrals to onsite food pantry or emergency food boxes if the onsite pantry is not open by 2024, 2) Pantry plus nutritious no-prep, ready-to-eat meals, or 3) Pantry plus $75 grocery vouchers for three-months. The study team will assess improvements in patient food security, diet quality, satisfaction, and wellbeing over time. Results of this pilot will inform the design of a food security response program for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Simmons cancer center
* Adults 18 years or older
* Ability to understand and willingness to provide informed consent
* Screens positive for food and/or nutrition insecurity
* No allergies or digestive diseases that could put participant at-risk of harm from consuming study foods (e.g., celiacs disease, dairy allergy, wheat allergy)

Exclusion Criteria:

* Not a patient at the Simmons cancer center
* Under 18 years of age
* Unable to provide informed consent
* Not wanting to participate
* Does not screen positive for food and/or nutrition insecurity
* Allergies or digestive diseases that could put participants at-risk of harm from consuming study foods (e.g., celiacs disease, dairy allergy, wheat allergy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Food security | 3-months
  6-item United States Department of Agriculture Food Security Screener (USDA); questionnaire; raw score 0-1-High or marginal food security, 2-4-Low food security, 5-6-Very low food security.

SECONDARY OUTCOMES:
Patient satisfaction | 3-months
  Satisfaction with clinical experience and interventions; two-items from the HCAHPS (Hospital Consumer Assessment of Healthcare Providers and Systems) Survey will be used to measure patient satisfaction with the clinical experience - items 21 & 22 on Overall Rating of Hospital (Q21) and Willingness to Recommend Hospital (Q22) - minimum = 0 (poorer quality care), maximum = 4 (higher quality care).
Patient wellbeing | 3-months
  The World Health Organisation-Five Well-Being Index (WHO-5), 5-items with 5 response options each, 0 to 25, 0 respresents worst possible quality of life and 25 represents best possible quality of life.

OTHER OUTCOMES:
Diet quality | 3-months
  Abbreviated Diet History Questionnaire III (DHQ-III) is a food frequency questionnaire (FFQ) that will be used to calculate a Healthy Eating Index score with a minimum value of 0 indicating poor dietary quality and a maximum value of 100 indicating high dietary quality.

CONTACTS AND LOCATIONS:
Overall Officials: Kelseanna Hollis-Hansen, PhD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be submitted to the PI 12 months after article publication. The data can be made accessible for up to 24 months for those who have access to secure data storage.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12-months after article publication, up to 24-months.
Access Criteria: Access to trial IPD can be requested by qualified researchers, and will be provided following review and approval of a research proposal that includes an analytic plan and a data sharing agreement. For more information or to submit a request, please contact the study team.

REFERENCES:
- [Background] Gany F, Melnic I, Wu M, Li Y, Finik J, Ramirez J, Blinder V, Kemeny M, Guevara E, Hwang C, Leng J. Food to Overcome Outcomes Disparities: A Randomized Controlled Trial of Food Insecurity Interventions to Improve Cancer Outcomes. J Clin Oncol. 2022 Nov 1;40(31):3603-3612. doi: 10.1200/JCO.21.02400. Epub 2022 Jun 16. PMID 35709430
- [Background] Berkowitz SA, Delahanty LM, Terranova J, Steiner B, Ruazol MP, Singh R, Shahid NN, Wexler DJ. Medically Tailored Meal Delivery for Diabetes Patients with Food Insecurity: a Randomized Cross-over Trial. J Gen Intern Med. 2019 Mar;34(3):396-404. doi: 10.1007/s11606-018-4716-z. Epub 2018 Nov 12. PMID 30421335